CLINICAL TRIAL: NCT02607839
Title: Regulation of Intestinal and Hepatic Lipoprotein Particle Production by Blood Glucose in Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Gary Lewis, Professor, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 12-5569-B
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: lipid handling by the gut and liver
MeSH Terms: interventions — Glucose; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- normal saline (Placebo Comparator): normal saline intravenous infusion
  Interventions: Biological: glucose or normal saline
- glucose (Active Comparator): glucose intravenous infusion
  Interventions: Biological: glucose or normal saline

INTERVENTIONS:
Biological: glucose or normal saline — 20% glucose solution or normal saline, intravenous infusion

SUMMARY:
The purpose of study is to examine whether raised blood glucose enhances lipid particle production independent of effects on gastric emptying and pancreatic/ gastrointestinal hormone production.

DETAILED DESCRIPTION:
This study will be performed on healthy, lean, non-diabetic males and females who will participate two studies each in random order, 4 to 6 weeks apart. Study A: lipoprotein turnover with intravenous infusion of normal saline. Study B: lipoprotein turnover i.v infusion of glucose. In both studies, subjects will drink a liquid formula every hour to remain in a constant fed state and will be under conditions of pancreatic clamp (with the infusion of hormones somatostatin, insulin, glucagon, growth hormone). Subjects will be blinded with regard to the treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18 to 60 years
2. Body mass index 20 kg/m2 to 27 kg/m2
3. Hemoglobin above 130g/L
4. Normal glucose tolerance in response to a 75g, 2-hr OGTT

Exclusion Criteria:

1. Subject has a history of hepatitis/hepatic disease that has been active within the previous two years.
2. Any subject with active bleeding, bleeding diathesis, clotting abnormalities or recent surgery (within past 1 month)
3. Any significant active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, renal (Cr > 1.5 mg/dL), genitourinary, hematological systems, or has severe uncontrolled treated or untreated hypertension (sitting diastolic BP > 100 or systolic > 180).
4. History of diabetes or OGTT indicative of diabetes or impaired glucose tolerance.
5. Any history of a MI or clinically significant, active, cardiovascular history including a history of arrhythmia's or conduction delays on ECG, unstable angina, or decompensated heart failure.
6. Any laboratory values: AST > 2x ULN; ALT > 2x ULN TSH > 6 mU/l
7. Current addiction to alcohol or substances of abuse as determined by the investigator.
8. Mental incapacity, unwillingness or language barrier precluding adequate understanding or cooperation
9. Taking any prescription or non-prescription medications at the time of the study
10. Having donated blood three months prior to and three months post study procedures
11. A pregnancy test will be performed 1 to 3 days prior to each study in all female subjects. Those who test positive for pregnancy will be excluded.
12. Known allergy, hypersensitivity or contraindication to receiving study medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Production of TRL-apoB48 between treatments | 10 hours

SECONDARY OUTCOMES:
Production of TRL-apoB100 between treatments | 10 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Tornto General Hospital, UHN, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Xiao C, Dash S, Morgantini C, Lewis GF. Intravenous Glucose Acutely Stimulates Intestinal Lipoprotein Secretion in Healthy Humans. Arterioscler Thromb Vasc Biol. 2016 Jul;36(7):1457-63. doi: 10.1161/ATVBAHA.115.307044. Epub 2016 May 5. PMID 27150393